CLINICAL TRIAL: NCT04857814
Title: Integrating Electronic Patient Reported Biometric Measures (ePReBMs) From ADAMM-RSM in Respiratory Diseases
Brief Title: Integrating Electronic Patient Reported Biometric Measures (ePReBMs) From Wearable Devices in Respiratory Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00097162
Record Dates: First submitted 2021-03-25; First posted 2021-04-23 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Progressive Fibrosing Interstitial Lung Disease; Lung Transplant; Cystic Fibrosis; Bronchiectasis; Pulmonary Tuberculosis
MeSH Terms: conditions — Cystic Fibrosis; Bronchiectasis; Tuberculosis, Pulmonary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Device (Experimental): All participants will wear the device to assist in determining the feasibility of wearing the device.
  Interventions: Device: ADAMM- RSM Device

INTERVENTIONS:
Device: ADAMM- RSM Device — All participants will wear the ADAMM- RSM device for a 6 month period

SUMMARY:
Lung diseases are one of the most common causes of emergency room visits. There are very few tools that are able to predict which patients will have a worsening or increasing severity of their condition. There are also limited ways to check the health of patients with respiratory conditions at home and during the time between medical appointments.

The ADAMM-RSMTM device records heart rate, breathing rate, temperature, cough and activity while wearing it. This study will test participants willingness to wear the device and perform ongoing monitoring to assess the possibility to predict the onset and increases in severity of their lung conditions.

DETAILED DESCRIPTION:
The project will aim to create the infrastructure to collect clinical data and participants reported biometric measures (ePReBMs) from wearable devices in a database, and to run a pilot phase with a limited number of participants. During this phase, the feasibility of a long-term (6 months) home monitoring of respiratory parameters with the wearable device ADAMM-RSM (Health Care Originals, Rochester, NY, USA) will be tested, in parallel with the standard of care, in a limited number of participants with progressive fibrosing interstitial disease (PF-ILD) including idiopathic pulmonary fibrosis (IPF), lung transplant, cystic fibrosis (CF) and bronchiectasis, and tuberculosis (TB). The study design will test the possibility to collect data from ADAMM-RSM: ideally, the participants should wear the ADAMM-RSM every day, for at least 8 hours. For the purpose of this study, the investigators will aim to collect data from the device for every participant at least 3 days per week, at least 8 hours per day, for a period of 6 months.

The duration of this study is estimated in 2 years, including the data analysis. The participants will be provided the due information about the study and they will sign a written consent before enrolment (a copy is attached to the application to the Research Ethics Office of the University of Alberta).

Every participant enrolled in the study will be asked to wear the ADAMM-RSM (Health Care Originals, Rochester, NY, USA) device every day for 6 months.

The wearable device includes a non-invasive biosensor and processor that is attached to the surface of the skin using an adhesive sticker. It is designed to measure physical activity, heart rate, respiration, skin temperature, and cough metrics using embedded audio transducers, thermistor, accelerometer, gyroscope, and magnetometer. It can be applied anywhere on the chest, with a single-use, changeable sticker. As such, the device is able to collect heart and respiratory rate, temperature and cough, and to correlate these parameters to rest, activity and intensity of activity for the duration of the battery (18 hours). After signing the informed consent, the participants will be instructed on how to apply and to remove the device on/from the chest, to use the device during the day, and to recharge it at night using its dedicated charger.

Every device is supplied with a unique anonymous identifier, and will transmit the data via Wi-Fi to a cloud secured database provided by Health Care Originals (Health Care Originals, Rochester, NY, USA). This database will be physically located in a server within the Canadian borders. The database will be moved to a secured server at the University of Alberta at the end of the study.

Potential registrations of speech during cough episodes are prevented by an integrated algorithm in the device, cleaning automatically any sound other than cough before transferring the data to the cloud server.

Local research coordinators will use a web-based portal to check the usage of the devices and that the devices are working properly. This portal does not include personal data of the participants but only the device identifier so matching back of actual patient to data stream will not occur on any of Healthcare Originals infrastructure.

A unique progressive study ID will be assigned to every participant entering the study. This ID will be coupled to the ADAMM-RSM identifier and it will be used in a separate database to collect clinical and follow-up data. The ID will be coupled to participants identifiers only in a third excel file, encrypted and protected with a password that will be accessible only to the study investigators.

The participants will be requested to fill 3 quality of life questionnaires (the King's Brief Interstitial Lung Disease questionnaire for PF-ILD or Saint George Respiratory Questionnaire for the other diagnoses, the Leicester Cough Questionnaire and the MRC dyspnea questionnaire for all the enrolled patients) at the time of enrolment, and after 3 and 6 months. The questionnaires will be used to compare responses at 3 and 6 months to the data generated from the device. Participants will be asked to return the device to the study site at the 6-month timepoint. Clinical data will be collected from the participant's chart if available at the baseline, 3, and 6 month timepoints as per the CRF's.

ELIGIBILITY:
Inclusion Criteria:

* Patients with PF-ILD (including IPF), lung transplant, CF, bronchiectasis or TB must meet all of the following criteria to be enrolled in the study:

  1. Male or female volunteers, at least 18 years of age at the time of screening visit;
  2. Fluent in English and able to follow the instructions to use the ADAMM-RSM™;
  3. Willing and cognitively able to sign informed consent

Exclusion Criteria:

* Patients must be excluded from participation in this study if any of the following criteria are met:

  1. Pregnancy;
  2. History of active (clinically significant) skin disorders;
  3. History of allergic response to silicones or adhesives;
  4. Subjects with electronic implants of any kind (e.g. pacemaker);
  5. Broken, damaged or irritated skin or rashes near the sensor application sites;
  6. Subjects who are physically or cognitively unable to normally perform activities of daily living, assessed at the discretion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Length of time wearing device (days) | 6 month duration per participant
  Total length of time participant wears device

SECONDARY OUTCOMES:
Prediction of respiratory exacerbations- Number of emergency room visits | 6 month duration per participant
  Explore the possibility to predict exacerbations/flares up of the respiratory condition of the patients
Prediction of respiratory exacerbations- Number of hospital admissions | 6 month duration per participant
  Explore the possibility to predict exacerbations/flares up of the respiratory condition of the patients

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Ferrara, MD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada